CLINICAL TRIAL: NCT03495388
Title: Pharmacogenetics and Pharmacokinetics of Oxycodone to Personalize Postoperative Pain Management Following Major Inpatient Surgery in Children
Brief Title: PG and PK of Oxycodone to Personalize Post-op Pain Management Following Surgery in Children
Status: Completed | Type: Observational
Sponsor: Senthil Sadhasivam (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY21070170; 7R01HD089458-02 (NIH)
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain; Opioid Dependence
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood is obtained and analyzed for genetic variations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Major Inpatient Surgeries: Children ages 8-17.9 undergoing pectus excavatum or idiopathic scoliosis spinal fusion at Riley Hospital for Children, who have consented to participate in an observational clinical study as approved by the IU IRB, protocol #1707525204.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Post-op pain management medication

SUMMARY:
Each year, in the U.S. alone, >6 million children undergo painful surgery; up to 50% of them experience significant and serious side effects with opioids and inadequate pain relief. Though 60% of this inter-individual variability in responses results from genetic variations, there is an almost complete lack of understanding of how specific genetic variability affects pain and of the adverse effects of opioids, especially in children. In this project the investigators will focus on oxycodone, a standard and preferred post-surgical oral analgesic in children

The purpose of this research is to study serious immediate and long-term clinical problems from both surgical pain and oxycodone use in children and adolescents to improve the safety and effectiveness of surgical pain relief.

The long-term goals are to improve the safety and effectiveness of surgical pain relief with opioids (a class of drugs/pain relievers) and to minimize the societal burden of disabling Chronic Persistent Surgical Pain (CPSP, which is pain that persists even after the expected healing time from surgery) and Opioid Dependence (OD) by preoperative risk predictions and personalized care with the right dose of the right pain medication for each child.

The overall objective is to determine the impact of risk factors on oxycodone's immediate and long-term negative postoperative outcomes and to personalize dosing in children undergoing outpatient and major inpatient surgery.

DETAILED DESCRIPTION:
Research procedures will include:

1. Pre-operative blood draw for genotyping candidate genes and exploratory genes and for future similar studies will be collected.
2. Standardized pre-, intra-, and post-operative care will be received by all participants. The study team will record medical history, demographic information, concomitant medications, vitals, pain scores, post-operative nausea and vomiting, and all medications given post-surgery for pain management throughout the participants in-patient stay.
3. Psychological questionnaires to assess pain, risk of developing OD and chronic pain, anxiety and depression will be administered pre-operatively, and 48-72 hours, 7-14 days, 2 months, 3 months, 6 months and 12 months post-operatively.
4. Quantitative Sensory Testing will be performed on up to 100 participants pre-operatively, and 48-72 hours,3 months and 12 months post-operatively.
5. Serial blood draws for oxycodone and methadone pharmacokinetic modeling will be collected from up to 200 participants. QTc measurements will also be recorded from pre- and post-operative EKGs for those participants in which methadone pharmacokinetic blood samples are collected.

ELIGIBILITY:
Inclusion Criteria:

* Boy and girls
* All races
* ASA physical status 1 and 2
* Scheduled for pectus excavatum repair or idiopathic scoliosis spinal fusion
* Children with OSA will be included but stratified as they have more opioid-related complications.

Exclusion Criteria:

* Allergy to oxycodone or methadone
* Developmental delay
* Neurological disorder
* Renal or liver disease
* Pre-operative pain requiring analgesics
* On inhibitors or inducers of CYP2D6 and CYP3A
* Cannot read, write and speak English fluently

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pectus excavatum repair and spinal fusions are two of the most painful surgery children and adolescents undergo. Therefore, the investigators aim to recruit 500 children and adolescents, 8-17.9 years of age, undergoing inpatient pectus excavatum repair or idiopathic scoliosis spinal fusions at Riley Hospital for Children.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Look at genetic factors predisposing children to immediate postoperative opioid-adverse effects (RD and PONV). | Immediately post-surgery during hospital stay and at home up to 1 year post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with children who experience RD, and PONV in the immediate post-surgical period (4 days) in the hospital and at home.
Look at genetic factors predisposing children to inadequate surgical pain relief with oxycodone. | Immediately post-surgery during hospital stay and at home up to 1 year post-surgery
  The investigators will look at specific CYP2D6, ABCB1, FAAH, OPRM1, and COMT variants to find correlations with children who experience poor pain relief in the immediate post-surgical period (4 days) in the hospital and at home.

SECONDARY OUTCOMES:
Look at the impact of CYP2D6 variants on oxycodone's clinical dosing in children to see if specific variants correlate with a need for lower or higher doses of analgesic. | Pre-operative to post-operative day 2
  The investigators will look at CYP2D6 variants to find correlations in oxycodone's PK variability and the need for dose adjustments that lead to desired clinical outcomes in children undergoing major inpatient surgeries.

OTHER OUTCOMES:
Look at genetic oxycodone-related perioperative and bio-psychological factors predisposing children to long-term adverse outcomes such as chronic persistant surgical pain and opioid dependence. | Pre-operative to 12 months post-operative
  The investigators will look at OPRM1 epigenetics and OPRM1, FAAH, GCH1, DRD2 variants to find correlations with chronic persistent surgical pain and opioid dependence up to 1 year post-surgery. Children will also be asked to complete psychological questionnaires pre-surgery, and at 4 time points post-surgery to assess psycho-psychological factors that may correlate with chronic persistent surgical pain or opioid dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, MPH, Principal Investigator — University of Pittsburgh, UPMC
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - UPMC Children's Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aruldhas BW, Quinney SK, Packiasabapathy S, Overholser BR, Raymond O, Sivam S, Sivam I, Velu S, Montelibano A, Sadhasivam S. Effects of oxycodone pharmacogenetics on postoperative analgesia and related clinical outcomes in children: a pilot prospective study. Pharmacogenomics. 2023 Mar;24(4):187-197. doi: 10.2217/pgs-2022-0149. Epub 2023 Mar 22. PMID 36946298
- [Derived] Packiasabapathy S, Aruldhas BW, Zhang P, Overholser BR, Quinney SK, Sadhasivam S. Novel associations between CYP2B6 polymorphisms, perioperative methadone metabolism and clinical outcomes in children. Pharmacogenomics. 2021 Jul;22(10):591-602. doi: 10.2217/pgs-2021-0039. Epub 2021 Jun 8. PMID 34100292
- [Derived] Sadhasivam S, Aruldhas BW, Packiasabapathy S, Overholser BR, Zhang P, Zang Y, Renschler JS, Fitzgerald RE, Quinney SK. A Novel Perioperative Multidose Methadone-Based Multimodal Analgesic Strategy in Children Achieved Safe and Low Analgesic Blood Methadone Levels Enabling Opioid-Sparing Sustained Analgesia With Minimal Adverse Effects. Anesth Analg. 2021 Aug 1;133(2):327-337. doi: 10.1213/ANE.0000000000005366. PMID 33481403